CLINICAL TRIAL: NCT01360411
Title: Tissue Characterisation Using Ultrasound Based Strain Imaging(Elastography)Examining Lesions in the Gastrointestinal Wall, Adjacent Lymph Nodes and Pancreatic Lesions
Brief Title: Tissue Characterisation by Endoscopic GI-elastography
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, Roald Flesland Havre, MD, Haukeland University Hospital
Other Study IDs: 17765
Record Dates: First submitted 2010-04-26; First posted 2011-05-25 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Disorder of Upper Gastrointestinal Tract; Pancreatic Nodule; Secondary and Unspecified Malignant Neoplasm of Retroperitoneal Lymph Nodes; Secondary Malignant Neoplasm of Lymph Node
Keywords: elastography; strain ratio; pancreas; GI wall lesions; lymph nodes
MeSH Terms: conditions — Neoplasm Metastasis; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples are stored as pathological slides in the diognostic biobank of Dep. of Pathology, Helse Bergen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pancreatic lesions: Any patient with a solid pancreatic lesion of unknown histology may be recruited. Cystic lesions are not included.
  Elastography findings are classified and compared to cytology or histology if the standard procedures or treatment provide this. In other cases the patients are being followed up conservatively.
- Intramural upper GI-lesions: Patients with intramural lesions discovered by endoscopy or other imaging modalities are recruited. Elastography findings are classified and compared to cytology or histology if the standard procedures or treatment provide this. In other cases the patients are being followed up conservatively.
- Lymph nodes: Patients with visible mediastinal lymph nodes or retroperitoneal lymph nodes in patients with inflammatory or malignant diseases are recruited. Elastography findings are classified and compared to cytology or histology if the standard procedures or treatment provide this. In other cases the patients are being followed up conservatively.

SUMMARY:
In this single centre study we study the use of endoscopic ultrasonography (EUS) combined with elastography in order to separate malignant tissue from benign tissue in and adjacent to the upper gastrointestinal tract.

DETAILED DESCRIPTION:
The purpose of this study is to use endoscopic ultrasonography (EUS) with strain based elastography to identify strain traits separating malignant from benign lesions. We are registering feasibility of endoscopic strain imaging and compare diagnostic accuracy of EUS + elastography with previous data on EUS alone.

Inclusion criteria:

* Group 1: Focal subepithelial lesions in esophageal, ventricular or duodenal wall discovered by endoscopy or other imaging modality.
* Group 2: Pancreatic lesion discovered by other imaging modality.
* Group 3: Mediastinal or retroperitoneal lymph node or tumor discovered by other imaging modality.

Histology of lesions should not be known at the time of examination. EUS elastography findings are evaluated shortly after the examination and categorised by different methods; categorical score, VAS, Strain Ratio. The result is then compared to histology or cytology results. Patients who do not undergo tissue sampling are followed up to discover disease progress.

ELIGIBILITY:
Inclusion Criteria:

* Solid focal lesions in pancreas or pancreatitis
* Intramural lesions in esophagus, ventricle or duodenum
* Lymph nodes or tumour > 1 cm in mediastinum or retroperitoneum accessible by EUS

Exclusion Criteria:

* Cystic pancreatic lesions
* Patients where the histology or cytology of the lesion in question is known at the time of examination

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients referred to EUS examination or relevant surgery at Haukeland University Hospital, bergen, Norway within the inclusion period (2007- January 2011).
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2007-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Malignant or benign lesion | Jan 2007 - September 2011 + 6 months( if no tissue sample)(4 years)
  Imaged lesions are sampled, surgically removed or followed up > 6 months to conclude on their nature. Images are evaluated, measured and categorised shortly after examination and compared to histological, cytological or follow up result. Elastography results do not interfere with surgical or oncological treatment planning in this study.

SECONDARY OUTCOMES:
Description of lesion elasticity | 2007- September 2011 (4 years)
  To identify softer and harder areas within and adjacent to focal lesions which could identify smooth surface, necrotic centre, regional fibrosis or regional cacncer.
Value of Strain Ratio measurements | 2007 - September 2011 (4 years)
  Strain ratio provides opportunity to compare strain in user selected areas of the elastogram. This is a semi-quantification of strain differences and may be useful for a better distinction between malignant ond non-malignant lesions.
Value of colour and pattern category | 2007 - September 2011 (4 years)
  Categorisation of images of lesions using a published categorising scheme and comparision to cytology, histology or follow up.
Value of a Visual Analog Scale for strain image categorisation | 2007 - September 2011 (4 years)
  Evaluation of the use of a simple 100 mm Visual analog scale to classify if lesion appears softer, equal to or harder than the surrounding tissue is useful for creating semiquantitative cut-off levels between malignant and benign lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Birger Nesje, MD, PhD, Study Director — University of Bergen; Roald F. Havre, MD, Principal Investigator — University of Bergen
Locations (1):
- Haukeland University Hospital/University of Bergen, Bergen, Norway

REFERENCES:
- [Background] Waage JE, Havre RF, Odegaard S, Leh S, Eide GE, Baatrup G. Endorectal elastography in the evaluation of rectal tumours. Colorectal Dis. 2011 Oct;13(10):1130-7. doi: 10.1111/j.1463-1318.2010.02440.x. PMID 21040360
- [Background] Havre RF, Elde E, Gilja OH, Odegaard S, Eide GE, Matre K, Nesje LB. Freehand real-time elastography: impact of scanning parameters on image quality and in vitro intra- and interobserver validations. Ultrasound Med Biol. 2008 Oct;34(10):1638-50. doi: 10.1016/j.ultrasmedbio.2008.03.009. Epub 2008 Jun 4. PMID 18524458
- [Background] Saftoiu A, Vilmann P, Gorunescu F, Janssen J, Hocke M, Larsen M, Iglesias-Garcia J, Arcidiacono P, Will U, Giovannini M, Dietrich C, Havre R, Gheorghe C, McKay C, Gheonea DI, Ciurea T; European EUS Elastography Multicentric Study Group. Accuracy of endoscopic ultrasound elastography used for differential diagnosis of focal pancreatic masses: a multicenter study. Endoscopy. 2011 Jul;43(7):596-603. doi: 10.1055/s-0030-1256314. Epub 2011 Mar 24. PMID 21437851
- [Background] Havre RF, Waage JR, Gilja OH, Odegaard S, Nesje LB. Real-Time Elastography: Strain Ratio Measurements Are Influenced by the Position of the Reference Area. Ultraschall Med. 2012 Dec;33(6):559-568. doi: 10.1055/s-0031-1273247. Epub 2011 Jun 10. PMID 21667433
- [Result] Saftoiu A, Vilmann P, Gorunescu F, Janssen J, Hocke M, Larsen M, Iglesias-Garcia J, Arcidiacono P, Will U, Giovannini M, Dietrich CF, Havre R, Gheorghe C, McKay C, Gheonea DI, Ciurea T; European EUS Elastography Multicentric Study Group. Efficacy of an artificial neural network-based approach to endoscopic ultrasound elastography in diagnosis of focal pancreatic masses. Clin Gastroenterol Hepatol. 2012 Jan;10(1):84-90.e1. doi: 10.1016/j.cgh.2011.09.014. Epub 2011 Oct 1. PMID 21963957